CLINICAL TRIAL: NCT05159726
Title: YOU MATTER: Using Video Education to Improve Patient Knowledge of Severe Maternal Morbidity (SMM) Warning Signs
Brief Title: Postpartum Video Education
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yale University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2000031817
Record Dates: First submitted 2021-12-08; First posted 2021-12-16 (Actual); Last update posted 2023-02-01 (Actual); Status verified 2023-01

CONDITIONS: Postpartum Hemorrhage; Postpartum Preeclampsia; Postpartum Sepsis; Postpartum Depression; Patient Empowerment; Patient Education; Postpartum Care
MeSH Terms: conditions — Postpartum Hemorrhage; Puerperal Infection; Depression, Postpartum; Patient Participation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Written Discharge Education + Video Education (Experimental): These patients will view a 12-minute educational video on SMM warning signs, in addition to the written discharge instructions provided by nursing staff. At the completion of the video, they will complete a post-video questionnaire to assess their knowledge on the covered topics.
  Interventions: Other: Video Education
- Written Discharge Education (No Intervention): They will receive the written discharge instructions provided by nursing staff and complete the post-discharge instruction questionnaire.

INTERVENTIONS:
Other: Video Education — 12-minute educational video covering postpartum topics of hemorrhage, infection, hypertension, and depression. Created by Cicatelli Associates Inc.
  Arms: Written Discharge Education + Video Education

SUMMARY:
This is a prospective, single-center, randomized control study to determine if video education at the time of postpartum discharge improves patient knowledge on the warning signs for the top three causes of severe maternal morbidity (infection, hemorrhage, and blood pressure disorders) in the first seven days following delivery. Participants will be randomized to written discharge education + video education (intervention) vs standard discharge education (control). They will complete a baseline questionnaire and a post-discharge education questionnaire during their postpartum stay to assess for knowledge improvement. The investigators hypothesize that video education will improve patient's knowledge of severe maternal morbidity warning signs.

DETAILED DESCRIPTION:
Prior to the day of postpartum discharge, a designated staff person will approach eligible patients and review the objectives of the study. If patients are willing to participate, they will complete a consent form and the baseline questionnaire. The baseline questionnaire will assess patient knowledge on postpartum hemorrhage, infection, hypertensive disorders of pregnancy, and depression.

Following delivery, patients will be randomized. Randomization will be done in a 1:1 allocation ratio between written discharge instructions + video education vs. written discharge instructions (standard of care at YNHH). A computer algorithm will assign participant based on random permuted blocks design with block size between 2-4. Each participant will have an assigned Study ID number that is linked to their random assignment. Group 1 will be the written discharge + video education group (intervention group). Group 2 will be the written discharge education (control group).

On the day of discharge, the nursing staff will provide discharge education based on their randomized group:

Group 1 will be the written discharge education + video education group (intervention group). These patients will view a 12-minute educational video on SMM warning signs, in addition to the written discharge instructions provided by nursing staff. At the completion of the video, they will complete a post-video questionnaire to assess their knowledge on the covered topics.

Group 2 will be the written discharge instruction group (control group). They will receive the written discharge instructions provided by nursing staff and complete the post-discharge instruction questionnaire.

Following discharge, patients will complete a post-discharge questionnaire to assess knowledge retention on the covered topics.

Patients' antepartum, delivery, and postpartum course will be reviewed until 1 year postpartum, including outpatient visits, emergency department visits, and any hospitalizations.

All subjects will be assigned a unique study ID code upon enrollment. Data will be collected from patients' medical records and from self-report. It will be recorded/stored in REDCap and on a Yale server accessible only to members of the research team. All data will be de-identified at the conclusion of chart review. Data analysts will have access to only de-identified information.

ELIGIBILITY:
Inclusion Criteria:

* Age >18 years
* Speaks English or Spanish
* Informed and written consent
* Delivered at Yale New Haven Hospital (YNHH)
* Received prenatal, and will receive postpartum, care through a YNHH-affiliated obstetric and/or midwifery practice

Exclusion Criteria:

* Patients who do not plan to receive postpartum care within the YNHH system
* Patients who experience an intrauterine fetal demise
* Patients who have a pregnancy with multiple severe congenital anomalies with an anticipated poor prognosis
* Patients who speak a primary language other than English or Spanish

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2022-07-05 (Actual); Primary Completion 2022-08-20 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
Change in baseline and post-education questionnaire score | Baseline, discharge (up to one week)
  Patients will complete a baseline and post-discharge education 15 item questionnaire that will assess knowledge on postpartum hemorrhage, infection, hypertensive disorders of pregnancy, and depression. The questionnaire will be scored 0-15 based on the number of correct responses. A lower score indicates lower knowledge, while a higher score indicates a better knowledge of the subject items. Outcome will be binary based on whether or not the patient improved their score between the two questionnaires.

SECONDARY OUTCOMES:
Change in post-education and post-discharge questionnaire score | 3-7 days
  Patients will complete a post-discharge questionnaire via email. The 15-item questionnaire will assess knowledge on postpartum hemorrhage, infection, hypertensive disorders of pregnancy, and depression. The questionnaire will be scored 0-15 based on the number of correct responses. A lower score indicates lower knowledge, while a higher score indicates a better knowledge of the subject items.
Compliance with Postpartum Care | 6 weeks
  The investigators will perform a retrospective chart review to determine if the study participant attended the 6 week postpartum visit
Healthcare utilization | 6 weeks
  The investigators will perform a retrospective chart review to determine number of phone call, clinic visits, urgent care and/or emergency room visits by each study participant
Patient satisfaction | Baseline, post-education
  Patients will rate their satisfaction with their knowledge and postpartum discharge on baseline and post-education questionnaires.

CONTACTS AND LOCATIONS:
Overall Officials: Heather Lipkind, MD, MPH, Principal Investigator — Yale University
Locations (1):
- Yale New Haven Hospital, New Haven, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Centers for Disease Control and Prevention. Pregnancy mortality surveillance system. Centers for Disease Control and Prevention, US Department of Health and Human Services; 2020. Accessed March 4, 2020. https://www.cdc.gov/reproductivehealth/maternal-mortality/pregnancy-mortality-surveillance-system.htm
- [Background] Petersen EE, Davis NL, Goodman D, Cox S, Mayes N, Johnston E, Syverson C, Seed K, Shapiro-Mendoza CK, Callaghan WM, Barfield W. Vital Signs: Pregnancy-Related Deaths, United States, 2011-2015, and Strategies for Prevention, 13 States, 2013-2017. MMWR Morb Mortal Wkly Rep. 2019 May 10;68(18):423-429. doi: 10.15585/mmwr.mm6818e1. PMID 31071074
- [Background] Centers for Disease Control and Prevention. (2019). Data Brief from 14 U.S. Maternal Mortality Review Committees, 2008-2017. Retrieved from https://www.cdc.gov/reproductivehealth/maternal-mortality/erase-mm/mmr-data-brief.html
- [Background] Human Resources & Services Administration. (2019). Maternal Morbidity & Mortality. Retrieved from https://www.hrsa.gov/maternal-mortality/index.html#about)
- [Background] Centers for Disease Control and Prevention. Severe Maternal Morbidity. Retrieved from https://www.cdc.gov/reproductivehealth/maternalinfanthealth/severematernalmorbidity.html
- [Background] Review to action, CDC Foundation. Capacity to review and prevent maternal deaths. report from nine maternal mortality review committees. 2018. http://reviewtoaction.org/Reportfrom_Nine_MMRCs.
- [Background] Krantz, T. E., et al. (2015). Computer graphic animation for intrauterine device contraceptive counseling in postpartum patients. Obstetrics and Gynecology 125: 68S.
- [Background] O'Dell, D. D., et al. (2019). A Quality Improvement Project- Standardizing Postpartum Discharge Instructions with an Educational Video. Obstetrics and Gynecology. Conference: 67th Annual Clinical and Scientific Meeting of the American College of Obstetricians and Gynecologists. Nashville, TN United States 133(SUPPL 1).
- [Background] O'Sullivan TA, Cooke J, McCafferty C, Giglia R. Online Video Instruction on Hand Expression of Colostrum in Pregnancy is an Effective Educational Tool. Nutrients. 2019 Apr 19;11(4):883. doi: 10.3390/nu11040883. PMID 31010174
- [Background] Wisely CE, Robbins CB, Stinnett S, Kim T, Vann RR, Gupta PK. Impact of Preoperative Video Education for Cataract Surgery on Patient Learning Outcomes. Clin Ophthalmol. 2020 May 20;14:1365-1371. doi: 10.2147/OPTH.S248080. eCollection 2020. PMID 32546944
- [Background] Che YJ, Gao YL, Jing J, Kuang Y, Zhang M. Effects of an Informational Video About Anesthesia on Pre- and Post-Elective Cesarean Section Anxiety and Recovery: A Randomized Controlled Trial. Med Sci Monit. 2020 Apr 8;26:e920428. doi: 10.12659/MSM.920428. PMID 32265432
- [Derived] White KJ, Tortal D, Callahan K, Eng K, Hyland M, Underwood E, Senter L, Leon-Martinez D, Son M, Lipkind H. Using a Patient Educational Video to Improve Knowledge of Maternal Mortality Warning Signs: A Randomized Controlled Trial. Obstet Gynecol. 2023 Nov 1;142(5):1139-1147. doi: 10.1097/AOG.0000000000005368. Epub 2023 Sep 13. PMID 37708502